CLINICAL TRIAL: NCT02938364
Title: Ear Plugs Versus Acupressure for Management of Severe Gag Reflex: A Randomized Clinical Trial
Brief Title: Ear Plugs Versus Acupressure for Management of Severe Gag Reflex
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riyadh Colleges of Dentistry and Pharmacy (Other)
Responsible Party: Principal Investigator, Mohammad Ramadan Rayyan, Assistant professor, Riyadh Colleges of Dentistry and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FUGRP/2016/115
Record Dates: First submitted 2016-10-17; First posted 2016-10-19 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Gagging
MeSH Terms: conditions — Gagging | interventions — Ear Protective Devices; Acupressure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Earplugs (Experimental): The participant will be asked to put plastic earplugs in both ears for 10 minutes and then the impression will be made while they are still on.
  Interventions: Other: Earplugs
- Acupressure (Experimental): The participant will be asked to wear sea bands on P6 points of both hand wrists for 10 minutes and then the impression will be made while they are still on.
  Interventions: Other: Acupressure
- Placebo (Placebo Comparator): The participant will be asked to wear non pressure bands on both hand wrists for 10 minutes and then the impression will be made while they are still on.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Earplugs — Plastic earplugs on both ears
  Arms: Earplugs
Other: Acupressure — Sea Bands put on the wrists of the participant to apply pressure on P6 points
  Arms: Acupressure
Other: Placebo — Non pressure bands put on the wrists of the participant
  Arms: Placebo

SUMMARY:
The aim of this study is to evaluate the efficacy of two proposed non-invasive techniques: the ear plug technique and acupressure on the P6 point in reducing gag reflex during impression making and to assess patient's experience in terms of comfort and satisfaction.

DETAILED DESCRIPTION:
The study will take place at the clinics of Riyadh Colleges of Dentistry and Pharmacy (RCsDP) in Riyadh, Saudi Arabia.

Patients, who on previous occasions have demonstrated difficulties in accepting the procedure of making impressions of maxillary teeth due to a severe gag reflex (GR) will be invited to participate in the study.

A Randomized single blinded clinical trial will be conducted on 30 participants who fulfill the inclusion criteria. Participants will be assigned to three separate groups. For each patient, two maxillary alginate impressions will be made; one before applying the proposed management technique and one after. Participants of Group EP (n=10) will be managed using earplugs while Group AC (n=10) will be managed using acupressure band and Group PL (n=10) will receive placebo management in forms of regular bands.

Informed consent will be obtained from all participants. All impressions will be made by one dentist that will be blinded to the gag reflex (GR) management techniques. The GR evaluation for all the participants will be performed by another calibrated dentist who is also blinded to the applied technique.

The severity of gag reflex will be assessed during making of the first impression using Dickinson & Fiske (2005) gagging severity index (GSI).

After 20 minutes of making the first impression, participants of Group EP will be asked to place the earplugs in and wait in the waiting room for 10 minutes. Then, the second impression will be made while the participant still has the earplugs on. Group AC will have acupressure technique via sea aid bands which will be placed on the P6 points of both hand wrists. Participants will be asked to wait in the waiting room for 10 minutes then the second impression will be made. PL Group will have the placebo management via placebo bands ( with no pressure points ) which will be placed on both hand wrists. Participants will also be asked to wait in the waiting room for 10 minutes then the second impression will be made. The effectiveness of the treatment will be assessed using Dickinson & Fiske (2005) gagging prevention index (GPI).

Participants will be asked to rate their discomfort during impression making using visual analogue scale (VAS).

ELIGIBILITY:
Inclusion Criteria:

* The individual is able to give informed consent.
* Patients with GR severity that are assigned to a gagging severity index (GSI) III-IV (for standardization of the baseline severity in between Groups).

Exclusion Criteria:

* Pregnant women
* Patients with Chronic heart diseases or cardiac pacemakers
* Patients with central or peripheral nervous system disorders
* Patients with oral lesions
* Patients with gastrointestinal disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-10-25 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Gagging severity index score | At the time of first impression which is made before applying the intervention method (baseline score) and again at the time of the second impression which is made after application of the intervention method by 10 minutes
  Gagging severity index (GSI) is a scale of gagging severity which ranges from 1 to 5 (very mild to very severe)

SECONDARY OUTCOMES:
Change from baseline Visual Analogue Scale scoring of patient's satisfaction during impression making | Directly after first impression which is made before applying the intervention (baseline score) and directly after the second impression which is made after application of the intervention method by 10 minutes
  The participant will be asked to score their judgment of the impression experience on a 0-10 scale where 0 refers to extremely pleasant and 10 refers to extremely unpleasant

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad R Rayyan, master, Principal Investigator — Riyadh Colleges of Dentistry and Pharmacy
Locations (1):
- Riyadh Colleges of Dentistry and Pharmacy, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided